CLINICAL TRIAL: NCT07011875
Title: The Effect of Physical Activity Levels on Dysmenorrhea Severity, Menstrual Symptoms, and Functional and Emotional Status in Women Diagnosed With Multiple Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Assistant Professor, Karabuk University
Other Study IDs: Multiple Sclerosis in Women
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Physical Activity; Dysmenorrhea; Emotional Disorder
Keywords: Multiple Sclerosis; Physical Activity Level; Dysmenorrhea Severity; Menstrual Symptom; Functional and Emotional Status
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with multiple sclerosis: Women diagnosed with multiple sclerosis by a neurologist

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, autoimmune disease that affects the central nervous system. It is more common in women, and hormonal factors are believed to play a role in its progression. The relapsing-remitting form of MS is particularly prevalent among women, leading to fluctuations in symptoms throughout the menstrual cycle.

One of the symptoms experienced during menstruation is dysmenorrhea, which can significantly impact quality of life due to severe pain and functional limitations. Dysmenorrhea is associated with both emotional and physical symptoms, and in women with MS, neurological symptoms may further intensify menstrual discomfort.

Physical activity is known to reduce inflammation and improve overall health. It has been shown to positively affect both MS symptoms and menstrual symptoms, including dysmenorrhea. However, research specifically examining the effects of physical activity on dysmenorrhea severity, menstrual symptoms, and emotional well-being in women with MS is limited.

This study aims to evaluate the impact of physical activity levels on dysmenorrhea severity, menstrual symptoms, and emotional well-being in women diagnosed with MS, addressing a gap in the literature and contributing to clinical practice.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, autoimmune, and demyelinating disease that causes damage to the white matter of the central nervous system. It is typically seen between the ages of 20 and 40. The incidence of MS is reported to be three times higher in women than in men. Although its etiology is not definitively known, it is thought that a combination of genetic predisposition and a non-genetic trigger-such as a virus, metabolism, or environmental factors-leads to recurring immune attacks on the central nervous system, resulting in a self-sustaining autoimmune disorder.

These factors, along with hormonal influences, contribute to the gender-related differences observed in MS. The main types of MS include relapsing-remitting, secondary progressive, primary progressive, and progressive-relapsing. The relapsing-remitting form is more common in women and is characterized by an earlier onset, more inflammatory lesions, and more frequent attacks. The higher prevalence of MS in women highlights the impact of hormonal factors on disease progression. Hormonal fluctuations throughout the menstrual cycle can cause variations in symptoms among women with MS. Some women with MS experience worsening symptoms before menstruation.

This worsening is most frequently reported in women with relapsing-remitting MS and is likely due to both new demyelinating plaques (exacerbation) and temporary symptom increases associated with previous plaques (pseudo-exacerbation). While the effects of hormonal fluctuations on MS are known, the overall impact of menstrual cycles on health should not be overlooked. The menstrual period is characterized by symptoms such as dysmenorrhea, which can negatively affect women's quality of life.

Dysmenorrhea is categorized into primary and secondary types. Primary dysmenorrhea is the most common form and is characterized by menstrual pain occurring before or during menstruation without any underlying pelvic disease. It typically begins 1-2 years after menarche or within 6-12 months and can persist until the age of 40. Dysmenorrhea is not limited to pain; it is also associated with emotional and physical symptoms such as irritability, depression, sleep disturbances, fatigue, decreased work performance, and functional limitations.

In women with MS, increased hormonal fluctuations may exacerbate existing neurological symptoms and intensify menstrual symptoms. This suggests that dysmenorrhea management in women with MS should be specifically evaluated. Physical activity is defined as any repetitive movement generated by skeletal muscles that results in an increased metabolic response compared to resting levels. Various studies have shown that regular physical activity is effective in reducing inflammation, supporting pain management, and improving psychological well-being.

In individuals with MS, the long-term immunomodulatory effects of physical activity are well known. Exercise has been shown to reduce inflammation and partially regulate neuroimmune parameters related to T-cell behavior. Similarly, physical activity has been reported to have a positive effect on menstrual symptoms such as dysmenorrhea. However, no studies have specifically investigated the impact of physical activity on dysmenorrhea severity, menstrual symptoms, and emotional status in women with MS.

Existing literature provides valuable insights into how physical activity affects disease symptoms in women with MS, but studies focusing on dysmenorrhea and menstrual symptoms are lacking. This study aims to fill this gap in the literature and contribute to clinical practice by evaluating the effects of physical activity levels on dysmenorrhea severity, menstrual symptoms, and functional and emotional status in women diagnosed with MS.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with multiple sclerosis by a neurologist

Aged between 18 and 55 years

Having an active menstrual cycle

Having a regular menstrual cycle (24-35 days)

No physical or cognitive impairment that prevents participation in exercise

Willingness to participate in the study

Exclusion Criteria:

* Postmenopausal status

Pregnancy or breastfeeding

Use of hormonal contraceptives or intrauterine devices

Use of medication that may affect dysmenorrhea

History of any gynecological surgery

Presence of pelvic pathology, pelvic inflammatory disease, endometriosis, or other conditions causing secondary dysmenorrhea

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study will include women with multiple sclerosis recruited from a patient association, focusing on those with active menstrual cycles to explore the relationship between physical activity and menstrual-related symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Baseline
  Participants will rate the intensity of menstrual pain using the Numerical Rating Scale from 0 (no pain) to 10 (worst pain imaginable). Only whole numbers will be used.
Functional and Emotional Impact of Dysmenorrhea | baseline
  This 14-item Likert-type scale evaluates the functional and emotional impact of dysmenorrhea. Each item is scored from 1 to 5. Higher scores indicate greater functional and emotional impairment.
International Physical Activity Questionnaire - Short Form | baseline
  Participants' physical activity levels during the last 7 days will be assessed using the IPAQ-Short Form. Results will be calculated in MET-minutes/week and categorized into three levels: inactive (<600 MET-min/week), low (600-3000 MET-min/week), and sufficient (>3000 MET-min/week).
Patient Determined Disease Steps | baseline
  Functional disability related to multiple sclerosis will be assessed using the PDDS, a patient-reported outcome scale ranging from 0 (normal) to 8 (bedridden). Higher scores indicate more severe disability.
Menstrual Symptom Questionnaire | baseline
  The Menstrual Symptom Questionnaire, consisting of 22 items rated on a 5-point Likert scale, will be used to assess somatic, emotional, and coping symptoms experienced during menstruation. Total scores range from 22 to 110, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Metehan YANA, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houtchens MK, Edwards NC, Schneider G, Stern K, Phillips AL. Pregnancy rates and outcomes in women with and without MS in the United States. Neurology. 2018 Oct 23;91(17):e1559-e1569. doi: 10.1212/WNL.0000000000006384. Epub 2018 Sep 28. PMID 30266889
- [Background] Guven Yorgun Y, Ozakbas S. Effect of hormonal changes on the neurological status in the menstrual cycle of patient with multiple sclerosis. Clin Neurol Neurosurg. 2019 Nov;186:105499. doi: 10.1016/j.clineuro.2019.105499. Epub 2019 Sep 10. PMID 31541863
- [Background] Harbo HF, Gold R, Tintore M. Sex and gender issues in multiple sclerosis. Ther Adv Neurol Disord. 2013 Jul;6(4):237-48. doi: 10.1177/1756285613488434. PMID 23858327
- [Background] Roeder HJ, Leira EC. Effects of the Menstrual Cycle on Neurological Disorders. Curr Neurol Neurosci Rep. 2021 May 10;21(7):34. doi: 10.1007/s11910-021-01115-0. PMID 33970361